CLINICAL TRIAL: NCT06927466
Title: A Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of B019 Injection in Subjects With Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceutical Group Biological Therapy Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B019-001
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B019 (Experimental)
  Interventions: Biological: B019

INTERVENTIONS:
Biological: B019 — B019： Intravenous infusion, 1.0×10^6 CAR T cell/kg-10.0×10^6 CAR T cell/kg

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of B019 in subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient himself/herself , and/or his/her legal guardian, agree to participate in the trial and sign the informed consent form；
2. Meet the diagnostic criteria for recurrent or refractory acute B cell lymphoblastic leukemia；
3. Documentation of CD19/CD22 tumor expression

3. Liver, kidney, lung and heart function meet requirements; 4. Expected survival >3 months; 5. Women of childbearing age and all post-adolescent male participants are willing to use highly effective contraceptive methods within 1 year after the infusion of B019 injection. At the same time, the subject should promise not to donate eggs or sperm for assisted reproduction for 1 year after the cell infusion.

-

Exclusion Criteria:

1. Active CNS involvement by malignancy；
2. Isolated extramedullary leukemia recurrence；
3. Subjects with ≥grade 2 acute or moderate to severe chronic graft-versus-host disease (GVHD) within 4 weeks prior to screening;
4. Has had treatment with any prior CAR-T therapy or other therapy abandoned in protocal.

4. Subjects who received therapy abandoned in protocal before PBMC (peripheral blood mononuclear cells) collection or before B019 injection; 5.Active other malignancy in 5 years. 6. Subjects who are positive for any of HBsAg, HBeAg, HBeAb, HBcAb, HCV-RNA, HIV EBV DNA, CMV DNA, HTLV-ab.

7. Other situations deemed inappropriate for participation in this study by the investigator.

-

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
(一) Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
The overall response rate (ORR) | 3 months
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Overall Survival (OS) | Approximately 2 years
  Determination of the overall survival times of all patients.
PK(Pharmacokinetics):Tmax | Approximately 2 years
  Time to peak plasma concentration (Tmax)
PK(Pharmacokinetics):Cmax | Approximately 2 years
  Maximum serum concentration(Cmax)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Peking University People's Hospital, Beijing
  - Jiangxi Province pediatric hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Children's Hospital of Soochow University, Suzhou
  - Tongji Hospital, Wuhan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou